CLINICAL TRIAL: NCT01625858
Title: Prospective Evaluation of Pediatric Supraglottic Airways in Anesthetized Children
Brief Title: Evaluation of Supraglottic Airway Devices in Children and Comparison to Historic Control
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: THLD-4-12
Record Dates: First submitted 2012-05-31; First posted 2012-06-21 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Evaluation of Success Rate; Airway Leak Pressure; Side Effects of LMA Supreme in Pediatric Patients Undergoing General Anesthesia
Keywords: LMA Supreme

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Supreme / other pediatric SGA: pediatric patients undergoing general anesthesia being treated with LMA Supreme or another pediatric supraglottic airway device

SUMMARY:
The supraglottic airway device LMA Supreme has recently been introduced for pediatric patients. The investigators will prospectively evaluate success rate and airway leak pressure in everyday's clinical pediatric anesthesia practice. Primary hypothesis is that the LMA Supreme has a leak pressure with a 95% confidence interval of 18-22cmH2O. Leak pressures will be compared to results from other pediatric supraglottic airway devices previously studied by the investigators group. Secondary Hypothesis: The primary success rate of the LMA-S is higher than 90%; therefore, performance is similar to the performance of the Ambu Aura Once™ and of the i-gel™. Study design: Prospective controlled observational cohort study.

In a second step, we will include more pediatric supraglottic airway devices. Each new arm will be handled exactly the same, assuming the same hypothesis being justified.

DETAILED DESCRIPTION:
The induction of anesthesia will follow the standard operating procedures of the pediatric anesthesia division at the children's hospital for the use of supraglottic airway devices. After loss of eyelash reflex and proper bag-mask ventilation provided, the SGA will be introduced into the mouth under standardized anesthesia to guarantee the same depth of anesthesia. This includes either propofol 2.5 mg/kg for older children, or sevoflurane inhalation in younger children at an end-tidal sevoflurane concentration of 6%. The time necessary to insert the airway device and the success rate will be recorded. We will also check at what airway pressure the SGA starts leaking. A fiberscope will be inserted through the airway port and through the gastric tube to obtain a view of the vocal cords and evaluate the position of the SGA. The gastric catheter will then be placed after insertion; the size will be according manufacturers' recommendations. After surgery, the SGA will be checked for evidence of mucosa lesions (blood stains on device). One day after surgery, the patient (and/or the parents) will be interviewed about sore throat, hoarseness, dysphagia, postoperative nausea and vomiting (PONV), rescue medication, pain, time of hospital discharge and any unscheduled re-hospitalization.

Before and during the operation, the following data will be recorded: Sex, age, weight, surgical procedure and duration, medications needed, cardiovascular parameter, depth of anesthesia. Secondary outcome data include:

* The insertion time necessary to airway device placement.
* Success rate of SGA device to ventilate patient
* Fiberscope view through the airway port on the glottis opening (1 full vision on the vocal cords - 4 no structure distinguishable)
* Fiberscope view through the airway gastric tube channel on the upper esophageal sphincter (rating 1-4)
* Placement of the gastric catheter (yes, no)
* Postoperative: Device will be checked for evidence of mucosa lesions (blood stains on device).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, ages 0-18 years, ASA physical status I-III, scheduled at the University Hospital of Bern for elective surgery under general anesthesia in supine position with planned operation time <4 hours and planned airway management including a supraglottic airway, written informed consent.

Exclusion Criteria:

* Exclusion criteria are high risk of aspiration of gastric content into the lungs, body mass index >35kg/m2, cervical spine disease, known difficult airway, upper respiratory tract symptoms in the previous 10 days, preoperative sore throat, poor dentition with high risk of damage, patients not speaking German or refusing to participate.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients of both genders, ages 0-18 years, ASA physical status I-III, scheduled at the University Hospital of Bern for elective surgery under general anesthesia in supine position with planned operation time <4 hours and planned airway management including a supraglottic airway.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Airway leak pressure | After 8 months
  Measured in cmH2O

SECONDARY OUTCOMES:
Number of LMA-S with primary success | After 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME, Study Chair — University Dept Anesthesiology and Pain Therapy, University of Berne, Switzerland
Locations (1):
- University Hospital Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Kleine-Brueggeney M, Gottfried A, Nabecker S, Greif R, Book M, Theiler L. Pediatric supraglottic airway devices in clinical practice: A prospective observational study. BMC Anesthesiol. 2017 Sep 2;17(1):119. doi: 10.1186/s12871-017-0403-6. PMID 28865448